CLINICAL TRIAL: NCT02705924
Title: Impact of a Psychoeducational Intervention on Expectations and Coping in Young Women (18-40 Years) Exposed to a High Familial Breast/Ovarian Cancer Risk
Brief Title: Impact of a Psychoeducational Intervention on Expectations and Coping in Young Women Exposed to a High HBOC Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 crisis prevents from organizing the last seminar
Sponsor: Centre Jean Perrin (Other)
Collaborators: Fondation de l'Avenir et la MASFIP, Paris - France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BRACAVENIR
Record Dates: First submitted 2016-03-02; First posted 2016-03-11 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducational intervention (Experimental): group participating to the first psychoeducational intervention: it consists in a week-end session in a SPA center including several conferences about HBOC familial risk, cancer prevention, prophylactic possibilities (surgery), recommendations about nutrition and physical activity a risk modulators, assisted medical procreation and embryo selection, social support...). Besides conferences, Moreno role games and group sharing are organized under the supervision of a psychotherapist.
  Interventions: Behavioral: psychoeducation
- Waiting list (Other): delayed intervention: group participating to the second psychoeducational intervention (6 months later). Intervention is same as in the intervention arm but it is delayed. Because questionnaires are completed before this second intervention in both arms and allocation to arms are randomized, it represents an adequate control group.
  Interventions: Behavioral: psychoeducation

INTERVENTIONS:
Behavioral: psychoeducation — Participants will attend conferences where experts present the state of the art in various domains:
  * Latest knowledge in oncogenetics
  * Recommendations and morbidity of prophylactic breast surgeries and annexectomy
  * Epidemiology of HBOC and comparative mortality risks with other syndromes/life habits
  * How to perform the periodic breast screening
  * Assisted medical procreation and embryo selection
  * Importance of nutrition and physical activity as risk modulator
  * Life habits: how one can increase or lower the cancer risk (tobacco, alcohol...)?
  * Description of the assistance program (GENAUV) to help counselees exposed to a high cancer risk follow their medical screening.
  The remaining time after this information, i.e. about half of the week-end, will comprise group activities, in particular role games (Moreno psychodrama approach) and group sharing under the supervision of a psychotherapist.

SUMMARY:
Young female counselees (18-40 years) belonging to HBOC families with a known mutation on BRCA-genes or not, receive a lot of information regarding their cancer risk. Information sources are numerous and sometimes contradictory. Unfortunately, these women face these issues at a key moment of there identity construction (self, relationship, sexuality) while they are not yet concerned by health prevention measures. A special psychoeducational intervention was designed to help these women to better cope with these difficulties.

Intervention consists in a week-end session in a thermal center (SPA) during which they will attend short conferences given by specialists (prevention measures, prophylactic surgery, assisted procreation, epidemiology...) and participate to role games and group sharing.

Intervention will be evaluated using self-questionnaires completed before intervention and during the following year.

DETAILED DESCRIPTION:
Background: Young women exposed to a high hereditary breast/ovaries cancer (HBOC) risk are particularly vulnerable: they are ignored by health prevention measures; they are embedded in a stream of contradictory information ( medicine, media, internet); they may feel concerned by surgical prevention issues at a key moment of there identity construction (self, relationship, sexuality). A special psychoeducational intervention was designed to help these women to better cope with these difficulties.

Methods/design: the study consists in a prospective randomized trial including childless young female counselees (18-40 years) of CCC Jean Perrin oncogenetics department, belonging to HBOC families either BRCA-mutated or not. They will be invited to attend a weekend group session in a SPA resort and participate to a series of short expert conferences and to focus group activities (group sharing, Moreno role game) supervised by a psychotherapist. Two sessions separated by a 6-month delay (waiting list) will enable us to evaluate the intervention effect, by comparing the evolution of questionnaires scores between inclusion and 6-month post-intervention. Main end-point is an increase of the Hert Hope Inventory of at least one standard deviation. Secondary endpoints investigate self-esteem, anxiety-trait, anxiety-state, ways of coping and quality of life. Participants will be randomized 1:1 to the first or the second session so that groups are comparable. Session will be cost-free for participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must belong to HBOC families,
* aged between 18 and 40 years
* Single or couple with a desire to have a child
* without any personal history of cancer.
* must have consulted at the oncogenetics department of the CCC Jean Perrin
* tested for a BRCA mutation.
* mutation carrier in case of a known familial BRCA mutation, else exposed to a high familial HBOC risk (Eisinger score ≥ 6 or Manchester score ≥ 16)
* must live in Auvergne region (middle France)
* signed an informed consent before inclusion.

Exclusion Criteria:

* pregnant women
* person who cannot answer questionnaires: language difficulties and/or cannot write in French correctly.
* no possible connection to our web-site
* psychiatric troubles and/or ongoing treatments preventing from a week-end stay in a SPA resort

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
changes in expectations measured using the Hert Hope Inventory questionnaire | changes of global score from baseline to 6-month post-intervention.
  Hert Hope Inventory global score [Herth, 1992, 2000] is used to evaluate expectations of participants. It contains only 12 simple proposals quoted using a 4-point Likert scale ranking from 1 = "strongly disagree" to 4 = "strongly agree". Its internal structure is composed of three dimensions: temporality and future, positive readiness and expectancy, and social/spiritual connectedness [Farran, 1995]. This questionnaire has been translated and validated in French by Lafrance [2013].

SECONDARY OUTCOMES:
Dimensions of coping evaluated by the Ways of Coping Checklist (WCC) [Folkman, 1980]. | inclusion - 6-month post-intervention - 1-year post-intervention
  The WCC French version contains 27 items quoted by Likert scales (answers within "no", "rather no", "rather yes", "yes"). Three specific dimensions are described:
  * the focus on the problem
  * the focus on emotions
  * the search for social support Dimensions will be used separately using their scores as no global score can be calculated (dimensions are divergent). This questionnaire has been validated in French in 1996 by Bruchon-Schweitzer et al.
Dimensions of perceived control measured using the Internal Powerful others and Chance scale (IPC) [Levenson, 1973]. | inclusion - 6-month post-intervention - 1-year post-intervention
  Perceived Control of IPC tests two locus of control: either in the self, or outside with two origins: fate/luck and "powerful others". Scores qualifying each locus of control will be used for statistics. This 24-item scale has been validated in French by Loas et al. [1994].
Level of Anxiety, either fundamental (as a trait of character) or superficial (depending on circumstances) evaluated by the State and Trait Anxiety Inventory (STAI A-B) [Spielberger, 1983] | inclusion - 6-month post-intervention - 1-year post-intervention
  The STAI A-B questionnaire evaluates anxiety in a way it cannot be confused with depressive syndrome. It comprises 40 items rated on a 4-point scale from "almost never" to "almost always". The 20 first ones evaluate the anxiety as a state, that is a labile/contextual form. The last 20 items estimate anxiety as a personality trait, independent of the environment. It has been translated and validated in French by Schweitzer & Paulhan [1990].
Score of the Self-Esteem Scale (SES) [Rosenberg, 1965] | inclusion - 6-month post-intervention - 1-year post-intervention
  It is a short 10-item questionnaire that evaluates the global self-worth by questioning positive and negative feelings about the self. The uni-dimensionality of the scale has been validated [Gray-Little, 1997]. The global score of the scale will be used as an indicator of self-esteem.
Subscales and global score of the WHO Quality of life questionnaire ( World Health Organization WHOQOL) [Harper, 1998]. | inclusion - 6-month post-intervention - 1-year post-intervention
  This questionnaire is worldwidely used. It contains four main dimensions: physical health, psychological, social relationships and environment. These dimensions have been confirmed in the French version by Leplège et al. [2000]. The global QoL score (means of subscales) will also be used for statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Yves-Jean BIGNON, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, Puy De Dome, France

IPD SHARING:
Plan to Share IPD: Undecided
answers to questionnaires

REFERENCES:
- [Background] Cousson-Gelie F, Cosnefroy O, Christophe V, Segrestan-Crouzet C, Merckaert I, Fournier E, Libert Y, Lafaye A, Razavi D. The Ways of Coping Checklist (WCC): validation in French-speaking cancer patients. J Health Psychol. 2010 Nov;15(8):1246-56. doi: 10.1177/1359105310364438. Epub 2010 Aug 27. PMID 20801945
- [Background] Bruchon-Schweitzer M, Cousson F, Quintard B, Nuissier J, Rascle N. French adaptation of the Ways of Coping Checklist. Percept Mot Skills. 1996 Aug;83(1):104-6. doi: 10.2466/pms.1996.83.1.104. PMID 8873181
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Folkman S, Lazarus RS. An analysis of coping in a middle-aged community sample. J Health Soc Behav. 1980 Sep;21(3):219-39. No abstract available. PMID 7410799
- [Background] Levenson H. Multidimensional locus of control in psychiatric patients. J Consult Clin Psychol. 1973 Dec;41(3):397-404. doi: 10.1037/h0035357. No abstract available. PMID 4803272
- [Background] Loas G, Dardennes R, Dhee-Perot P, Leclerc V, Fremaux D. [Operationalization of the "locus of control" concept: translation and first validation study of the Levenson control scale (IPC: the internal powerful others and chance scale)]. Ann Med Psychol (Paris). 1994 Aug-Sep;152(7):466-9. French. PMID 7978779
- [Background] Power M, Harper A, Bullinger M. The World Health Organization WHOQOL-100: tests of the universality of Quality of Life in 15 different cultural groups worldwide. Health Psychol. 1999 Sep;18(5):495-505. doi: 10.1037//0278-6133.18.5.495. PMID 10519466
- [Background] Leplege A, Reveillere C, Ecosse E, Caria A, Riviere H. [Psychometric properties of a new instrument for evaluating quality of life, the WHOQOL-26, in a population of patients with neuromuscular diseases]. Encephale. 2000 Sep-Oct;26(5):13-22. French. PMID 11192800
- [Result] Herth K. Enhancing hope in people with a first recurrence of cancer. J Adv Nurs. 2000 Dec;32(6):1431-41. doi: 10.1046/j.1365-2648.2000.01619.x. PMID 11136411
- [Derived] Kwiatkowski F, Gay-Bellile M, Dessenne P, Laquet C, Boussion V, Beguinot M, Petit MF, Gremeau AS, Verlet C, Chaptal C, Broult M, Jouvency S, Duclos M, Bignon YJ. BRACAVENIR: an observational study of expectations and coping in young women with high hereditary risk of breast and ovarian cancer. Hered Cancer Clin Pract. 2019 Feb 27;17:7. doi: 10.1186/s13053-019-0107-7. eCollection 2019. PMID 30858899
- [Derived] Kwiatkowski F, Dessenne P, Laquet C, Daures JP, Gay-Bellile M, Bignon YJ. BRACAVENIR - impact of a psychoeducational intervention on expectations and coping in young women (aged 18-30 years) exposed to a high familial breast/ovarian cancer risk: study protocol for a randomized controlled trial. Trials. 2016 Oct 21;17(1):509. doi: 10.1186/s13063-016-1642-4. PMID 27769293